CLINICAL TRIAL: NCT05460091
Title: Effect of High-Frequency Vibration on Periodontal Tooth Mobility
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00102774
Record Dates: First submitted 2022-07-07; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Tooth Mobility
Keywords: vibration; high-frequency; high frequency; effect
MeSH Terms: conditions — Tooth Mobility

STUDY DESIGN:
Intervention Model Description: Pilot RCT. We had a test group and a control group
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Graduate student and PI were double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Sham Comparator): Control group - sham Ptech device(does not vibrate)
  Interventions: Device: PTech Sham Device
- Test group (Active Comparator): Test group - active Ptech device (High-Frequency Vibrational device)
  Interventions: Device: PTech Device

INTERVENTIONS:
Device: PTech Device — High-frequency vibration device used on regular basis in orthodontics
  Arms: Test group
Device: PTech Sham Device — sham device (does not vibrate)
  Arms: Control Group

SUMMARY:
According to the CDC, approximately 47% of the population suffers from moderate or severe periodontitis. A byproduct of periodontal disease is loss of the alveolar bone surrounding the natural tooth root as well as around the dental implant in cases of peri-implantitis, and if allowed to proceed far enough, can cause mobility and eventual loss of the tooth or implant. Traditional and time-tested methods of treating periodontitis involve a meticulous mechanical cleaning of the root surfaces to remove the causing factors, both above and below the gumline. This reduction or elimination of the etiologic factors that trigger the pathologic and damaging immune response is very effective at reducing the inflammation. High Frequency Vibration (VPro+), when used as an adjunctive therapy following traditional treatment for periodontitis where the chronic inflammation has been lowered, controlled or eliminated has the potential to enhance the mechanical properties of the bone by increasing bone density by way of a low-risk, non-invasive, self-applied therapy that is patient-friendly and affordable. Improvement in bone density can translate clinically to lowering of tooth mobility, and lessening the chance of orthodontic relapse after orthodontic therapy. It is further hypothesized that, if conducted in an environment of low or nonexistent periodontal inflammation, VPro+ therapy may also contribute to enhanced the degree of bone fill after healing of angular periodontal bone defects and low-grade furcation involvements, and as thus may turn out to be a less invasive and more affordable option to periodontal bone grafting surgery, the current standard of care for those particular situations. The goal is to conduct a randomized clinical trial using patients in our graduate periodontology program to test the efficacy of high frequency vibration in improvement of tooth mobility and other periodontal indices in test group versus control group.

DETAILED DESCRIPTION:
Background Bio stimulation of hard and soft tissue to enhance or accelerate healing is an exciting area of inquiry with the potential to have broad clinical application in periodontics. The external application of energy in the form of light (e.g. Lasers or broad-spectrum light) (1) or mechanical waves (ultrasonic or high-frequency vibration) (2),(3) has shown efficacy in creating clinical changes in hard and soft tissue that can be very positive and beneficial or the contrary, depending on the application and the existing initial conditions present. According to the CDC, approximately 47% of the population suffers from moderate or severe periodontitis. (4) This chronic disease is a systemic disease that is fundamentally connected to other diseases of inflammation, including diabetes, arthritis, Alzheimer's Disease, and heart disease(5) and is, therefore, a disease that should not be taken lightly. A by-product of periodontal disease is the loss of the alveolar bone surrounding the natural tooth root as well as around the dental implant in cases of peri-implantitis, and if allowed to proceed far enough can cause mobility and eventual loss of the tooth or dental implant. The chronic inflammatory process results in the destruction of both hard and soft tissues and is triggered in the susceptible host by microbial biofilm and mineralized biofilm (i.e. calculus).

Traditional and time-tested methods of treating periodontitis involve a meticulous mechanical cleaning of the root surfaces to remove the causing factors, both above and below the gum line. This reduction or elimination of the etiologic factors that trigger the pathologic and damaging immune response is very effective at reducing inflammation. High-Frequency Vibration (VPro+), when used as an adjunctive therapy following traditional treatment for periodontitis wherein the chronic inflammation has been lowered, controlled, or eliminated has the potential to enhance the mechanical properties of the bone by increasing bone density (3) by way of a low-risk, non-invasive, self-applied therapy that is patient-friendly and affordable. Improvement in bone density can translate clinically to lowering (i.e. improvement) of tooth mobility and lessening the chance of orthodontic relapse after orthodontic therapy. It is further hypothesized that, if conducted in an environment of low or nonexistent periodontal inflammation, VPro+ therapy may also contribute to enhancing the degree of bone fill after healing of angular periodontal bone defects and low-grade furcation involvements, and as thus may turn out to be a less invasive and more affordable option to periodontal bone grafting surgery, the current standard of care for those particular situations.

Tissue Response to VPro+ Application in areas of Inflammation It is clear from previous research into the use of the VPro+ to accelerate and enhance orthodontic therapy that the cellular tissue response in areas of inflammation is essentially the opposite to that which occurs in areas of no inflammation. (3) Again, whether the response is beneficial depends on the intended application at hand. VPro+ therapy in areas of inflammation caused by orthodontic tooth movement forces stimulates osteoclastic activity to accelerate the resorption of bone, making the bone "softer" and thus allowing for more rapid tooth movement through these softer areas. On the contrary, when considering periodontitis, it is critical to understand that the inflammation must first be lowered and controlled so that the tissue response is anabolic, not catabolic. Our goal in periodontal therapy is to preserve, regenerate and strengthen the periodontal tissues, including the bone. So, a mandatory precursor therapy to using the VPro+ in cases of periodontitis is to first perform periodontal therapy and demonstrate and document a reduction or elimination of chronic inflammation by way of a Re-Evaluation Examination.

Expected result of this study We expect that VPro+ will safely enhance the condition of the periodontal tissues around the teeth in periodontal patients in a periodontal recall program and that this enhancement will improve the long-term prognoses of the teeth.

Study design This randomized, single blind clinical trial will enroll from 10-20 subjects from an established graduate periodontology program who have previously been treated for periodontal disease and are now in a periodontal recall program. These patients will be randomized between the two groups. The evaluator examining the patients will be blinded to the group assignment as the coding will be kept separate from the clinical patient record. The subjects, however, will be aware of whether they are in the treatment or no-treatment control group.

Specific Aims of the study:

This clinical trial aims to answer these questions:

1. Will the vibration produced by the VPro+ device improve (i.e. lessen) the mobility of periodontally compromised teeth for periodontal patients in a periodontal recall program?
2. Will the vibration produced by the VPro+ device improve the periodontal condition around teeth as measured by the standard periodontal indices in periodontal patients who are in a periodontal recall program?
3. Will the vibration produced by the VPro+ device improve the appearance of angular bone defects on routine radiographs (i.e. give the appearance of partial or complete fill of the bone defect) in periodontal patients in a periodontal recall program?
4. Will the vibration produced by the VPro+ device improve (i.e. increase) the bone density as measured by CBCT analysis in periodontal patients in a periodontal recall program? Study Groups

To address this specific aim, patient will be divided into 2 groups:

Group 1 (Treatment) This group will use the VPro+ device for 5 minutes every night for 3 months Group 2 (No Treatment) This group will be given a sham VPro+ device and thus serve as the control group.

Methods and procedures This is a randomized, single blinded clinical trial. The subjects will be patients with a history of treated periodontal disease that are currently in and compliant with a periodontal recall program in an established periodontal specialty practice. The subjects will be randomized between 2 groups. Group 1 is the treatment group and will receive the VPro+ device to use 5 minutes per night for 3 months. Group 2 is the no-treatment (control) group that will have access to the sham VPro+ device. Patient will be asked to bite comfortably on VPro+ for a total of 5 minutes per day, preferably just before bedtime. Compliance will be collected from the VPro+ using the Propel Application on the subjects' smartphone.

Data collection, data analysis and monitoring A designated clinical study coordinator will be assigned by the Principal Investigator. Good Clinical Practices (GCP) will be implemented for this study. The designee will review the Case Report Forms (CRF) for completeness and assess them for any product complaints, potential adverse events and/or medical device reports per the Health Canada regulations. Any missing entries in the CRFs will be brought to the Investigator or study coordinator's attention for correction.

Potential Benefits to the Subject In patients with periodontal disease and bone loss that have already been treated by traditional methods, we anticipate that the bone density and mechanical properties of the bone may increase (i.e. improve) in patients receiving HFV therapy. This can have the effect of lowering the mobility of some of the teeth. Even so, the subject may not get any benefit from being in this research study. This study may help people in the future who are in periodontal recall programs. Subjects (i.e. patients) who complete the study will not be charged for any of the care delivered during the study. Once the study is over, patients will go back on their normal periodontal recall program.

ELIGIBILITY:
Inclusion Criteria:

1. Overall health must be either ASA Classification I or II. (ASA I: A normal healthy patient; ASA II: A patient with mild systemic disease) (Doyle, Goyal, & EH, 2022),
2. Patient must have a recent history of treated periodontal disease and currently be compliant with a periodontal recall maintenance program supervised by a periodontal specialist,
3. Patient age must be between 30 and 85 years,
4. No gender or ethnic restrictions,
5. Patient must have at least one tooth with Miller's Class I mobility,
6. Patients should have posterior dentition such that they can firmly hold the vibrating device, this likely implies the presence of two or more posterior teeth in all four quadrants.

Exclusion Criteria:

1. Patients on medication that could affect the level of inflammation, such as chronic antibiotics, phenytoin, cyclosporine, anti-inflammatory drugs, systemic corticosteroids, or calcium channel blockers,
2. Periodontal recall patients who have a history of non-compliance with the recommended recall interval (usually three to four months),
3. Pregnant women,
4. Uncontrolled diabetes,
5. Smoking,
6. Subjects with current caries activity,
7. Vulnerable subjects as per the Research Ethics Office or HREB definitions.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Tooth Mobility | 3 months of intervention after use of device for 5 minutes per night
  Change in tooth mobility as denoted by Periotest value or Miller's grade of mobility

SECONDARY OUTCOMES:
Bone mineral density (BMD) | 3 months of intervention after use of device for 5 minutes per night
  Change in BMD as denoted by gray-scale values measured in Hounsfield units

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, Oral health Clinic, University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carroll JD, Milward MR, Cooper PR, Hadis M, Palin WM. Developments in low level light therapy (LLLT) for dentistry. Dent Mater. 2014 May;30(5):465-75. doi: 10.1016/j.dental.2014.02.006. Epub 2014 Mar 21. PMID 24656472
- [Background] El-Bialy T, Farouk K, Carlyle TD, Wiltshire W, Drummond R, Dumore T, Knowlton K, Tompson B. Effect of Low Intensity Pulsed Ultrasound (LIPUS) on Tooth Movement and Root Resorption: A Prospective Multi-Center Randomized Controlled Trial. J Clin Med. 2020 Mar 16;9(3):804. doi: 10.3390/jcm9030804. PMID 32188053
- [Background] Alikhani M, Alansari S, Hamidaddin MA, Sangsuwon C, Alyami B, Thirumoorthy SN, Oliveira SM, Nervina JM, Teixeira CC. Vibration paradox in orthodontics: Anabolic and catabolic effects. PLoS One. 2018 May 7;13(5):e0196540. doi: 10.1371/journal.pone.0196540. eCollection 2018. PMID 29734391
- [Background] Eke PI, Dye BA, Wei L, Thornton-Evans GO, Genco RJ; CDC Periodontal Disease Surveillance workgroup: James Beck (University of North Carolina, Chapel Hill, USA), Gordon Douglass (Past President, American Academy of Periodontology), Roy Page (University of Washin. Prevalence of periodontitis in adults in the United States: 2009 and 2010. J Dent Res. 2012 Oct;91(10):914-20. doi: 10.1177/0022034512457373. Epub 2012 Aug 30. PMID 22935673
- [Background] Friedewald VE, Kornman KS, Beck JD, Genco R, Goldfine A, Libby P, Offenbacher S, Ridker PM, Van Dyke TE, Roberts WC; American Journal of Cardiology; Journal of Periodontology. The American Journal of Cardiology and Journal of Periodontology editors' consensus: periodontitis and atherosclerotic cardiovascular disease. J Periodontol. 2009 Jul;80(7):1021-32. doi: 10.1902/jop.2009.097001. PMID 19563277